CLINICAL TRIAL: NCT05933577
Title: A Phase 3, Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled Clinical Study of Adjuvant V940 (mRNA-4157) Plus Pembrolizumab Versus Adjuvant Placebo Plus Pembrolizumab in Participants With High-Risk Stage II-IV Melanoma (INTerpath-001)
Brief Title: A Clinical Study of Intismeran Autogene (V940) Plus Pembrolizumab in People With High-Risk Melanoma (V940-001)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V940-001; V940-001 (Other: MSD); 2023-503652-27-00 (Registry Identifier: EU CT); jRCT2041230169 (Registry Identifier: jRCT); U1111-1287-6366 (Registry Identifier: UTN)
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Saline Solution; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intismeran autogene + Pembrolizumab (Experimental): Participants receive up to 9 doses of intismeran autogene via an intramuscular (IM) injection (every 3 weeks) plus up to 9 doses of pembrolizumab via an intravenous (IV) infusion (once every 6 weeks) until disease recurrence or unacceptable toxicity, or for a total treatment duration of up to approximately 56 weeks, whichever is sooner.
  Interventions: Biological: Intismeran autogene; Biological: Pembrolizumab
- Placebo + Pembrolizumab (Active Comparator): Participants receive up to 9 doses of dose matched placebo to intismeran autogene via an IM injection (every 3 weeks) plus up to 9 doses of pembrolizumab via an IV infusion (once every 6 weeks) until disease recurrence or unacceptable toxicity, or for a total treatment duration of up to approximately 56 weeks, whichever is sooner.
  Interventions: Biological: Pembrolizumab; Other: Placebo

INTERVENTIONS:
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; Individualized neoantigen therapy; V940
  Arms: Intismeran autogene + Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®
Other: Placebo — IM injection
  Other Names: Normal saline; Dextrose
  Arms: Placebo + Pembrolizumab

SUMMARY:
The purpose of this study is to learn if intismeran autogene which is an individualized neoantigen therapy (INT; formerly, called messenger ribonucleic acid [mRNA]-4157) with pembrolizumab (MK-3475) is safe and prevents cancer from returning in people with high-risk melanoma. Researchers want to know if intismeran autogene with pembrolizumab is better than receiving pembrolizumab alone at preventing the cancer from returning.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has surgically resected and histologically/pathologically confirmed diagnosis of Stage IIB or IIC, III, or IV cutaneous melanoma
* Has not received any prior systemic therapy for their melanoma beyond surgical resection
* No more than 13 weeks have passed between final surgical resection that rendered the participant disease-free and the first dose of pembrolizumab
* Is disease free at the time of providing documented consent for the study
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has ocular or mucosal melanoma
* Has cancer that has spread to other parts of the body and cannot be removed with surgery
* Has heart failure within the past 6 months
* Has received prior cancer therapy or another cancer vaccine
* Has another known cancer that that has spread to other parts of the body or has required treatment within the past 3 years
* Has severe reaction to study medications or any of their substance used to prepare a drug
* Have not recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2029-10-26 (Estimated); Study Completion 2030-09-26 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to approximately 74 months
  RFS is defined as the length of time from when the participant starts the study until either the cancer comes back, or the cancer spreads as assessed by the investigator, or death due to any cause.

SECONDARY OUTCOMES:
Distant Metastasis-Free Survival (DMFS) | Up to approximately 85 months
  DMFS is the length of time from when the participant starts the study until either the cancer spreads from where it started to other parts of the body as assessed by the investigator, or death due to any cause.
Overall-Survival (OS) | Up to approximately 85 months
  OS is the length of time that people are alive after joining the study.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 68 weeks
  An AE is a health problem that happens or worsens during a study. Number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 56 weeks
  An AE is a health problem that happens or worsens during a study. Number of participants who discontinue study treatment will be reported.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" will be scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better overall health status. Per protocol, the change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better level of physical functioning. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Role Functioning (Items 6 and 7) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a more impaired level of role functioning. Change from baseline in the role functioning (EORTC QLQ-C30 Items 6-7) combined score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (165):
- United States (34):
  - Highlands Oncology Group ( Site 1943), Springdale, Arkansas
  - UCLA Hematology/Oncology - Westwood (Building 100) ( Site 1918), Los Angeles, California
  - UCSF Medical Center at Mission Bay ( Site 1929), San Francisco, California
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 1933), New Haven, Connecticut
  - Orlando Health Cancer Institute ( Site 1937), Orlando, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center ( Site 1945), Tampa, Florida
  - Winship Cancer Institute of Emory University ( Site 1940), Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 1950), Marietta, Georgia
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 1935), Iowa City, Iowa
  - Johns Hopkins Hospital-Sidney Kimmel Comprehensive Cancer Center - Melanoma ( Site 1912), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 1927), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 1957), Boston, Massachusetts
  - Dana-Farber Cancer Institute ( Site 1956), Boston, Massachusetts
  - University of Michigan ( Site 1915), Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 1932), Grand Rapids, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1944), Hackensack, New Jersey
  - Atlantic Health System ( Site 1925), Morristown, New Jersey
  - Valley Health Systems - Ridgewood Campus ( Site 1947), Ridgewood, New Jersey
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 1958), Mineola, New York
  - NYU Langone Health-Perlmutter Cancer Center ( Site 1917), New York, New York
  - Columbia University Irving Medical Center-CUIMC Herbert Irving Comprehensive Cancer Center Clinical ( Site 1908), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1914), New York, New York
  - University of North Carolina Medical Center-Lineberger Comprehensive Cancer Center ( Site 1949), Chapel Hill, North Carolina
  - Duke Cancer Institute ( Site 1911), Durham, North Carolina
  - Hospital of the University of Pennsylvania Perelman Center for Advanced Medicine ( Site 1905), Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center ( Site 1909), Pittsburgh, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center ( Site 1934), Charleston, South Carolina
  - Sanford Cancer Center ( Site 1951), Sioux Falls, South Dakota
  - SCRI Oncology Partners ( Site 1910), Nashville, Tennessee
  - Texas Oncology - Austin ( Site 1903), Austin, Texas
  - Texas Oncology - Dallas (Sammons) ( Site 1902), Dallas, Texas
  - University of Texas MD Anderson Cancer Center ( Site 1920), Houston, Texas
  - Inova Schar Cancer Institute ( Site 1900), Fairfax, Virginia
  - Fred Hutchinson Cancer Center ( Site 1901), Seattle, Washington
- Argentina (6):
  - Clinica Adventista Belgrano-Oncology ( Site 2204), Caba., Buenos Aires
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 2202), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 2203), Buenos Aires, Buenos Aires F.D.
  - Centro Privado de RMI Río Cuarto S.A. II ( Site 2201), Río Cuarto, Córdoba Province
  - Hospital Aleman ( Site 2200), Buenos Aires
  - Sanatorio Finochietto ( Site 2205), Buenos Aires
- Australia (6):
  - Westmead Hospital ( Site 1001), Westmead, New South Wales
  - Melanoma Institute Australia-Clinical Trials Unit ( Site 1000), Wollstonecraft, New South Wales
  - Princess Alexandra Hospital ( Site 1003), Brisbane, Queensland
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 1005), Melbourne, Victoria
  - Paula Fox Melanoma & Cancer Centre ( Site 1004), Melbourne, Victoria
  - One Clinical Research ( Site 1002), Nedlands, Western Australia
- Belgium (5):
  - UZ Brussel-Medische oncologie ( Site 3405), Brussels, Bruxelles-Capitale, Region de
  - Ziekenhuis Oost-Limburg, Campus St.-Jan ( Site 3402), Genk, Limburg
  - UZ Gent ( Site 3403), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 3400), Leuven, Vlaams-Brabant
  - AZ Groeninge Campus Kennedylaan-Oncology ( Site 3401), Kortrijk, West-Vlaanderen
- Brazil (5):
  - Centro Avançado de Tratamento Oncológico- CENANTRON ( Site 2303), Belo Horizonte, Minas Gerais
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 2302), Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição ( Site 2309), Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Câncer - INCA-Pesquisa Clinica HC II ( Site 2305), Rio de Janeiro
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 2300), São Paulo
- Canada (7):
  - Cross Cancer Institute ( Site 1104), Edmonton, Alberta
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 1106), Vancouver, British Columbia
  - William Osler Health System ( Site 1105), Brampton, Ontario
  - Sunnybrook Research Institute ( Site 1103), Toronto, Ontario
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 1102), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal-Unité de Recherche Clinique en Oncologie et Hématolo ( Site 1100), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université L-Hemato-Oncology ( Site 1101), Québec, Quebec
- Chile (3):
  - FALP-UIDO ( Site 2400), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo-Hemato-Oncology ( Site 2402), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2401), Santiago, Region M. de Santiago
- Colombia (4):
  - Clinica Somer-Unidad de Investigacion y Docencia ( Site 2506), Rionegro, Antioquia
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 2500), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 2503), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 2505), Cali, Valle del Cauca Department
- Denmark (3):
  - Herlev and Gentofte Hospital ( Site 3301), Copenhagen, Capital Region
  - Aalborg Universitetshospital, Syd ( Site 3302), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 3300), Odense C, Region Syddanmark
- France (11):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet-Dermatology Department ( Site 1211), Nice, Alpes-Maritimes
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Ti-Service de Dermatologie et Cancérologi ( Site 1203), Marseille, Bouches-du-Rhone
  - Centre Georges François Leclerc ( Site 1210), Dijon, Cote-d Or
  - CHU Besançon ( Site 1209), Besançon, Doubs
  - CHU de Bordeaux Hop St ANDRE-Service de Dermatologie ( Site 1204), Bordeaux, Gironde
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 1206), Rennes, Ille-et-Vilaine
  - Hopital Claude Huriez - CHU de Lille ( Site 1207), Lille, Nord
  - centre hospitalier lyon sud-Service de dermatologie ( Site 1202), Pierre-Bénite, Rhone
  - CHU d'Amiens-Picardie - Hôpital Sud-Dermatologie ( Site 1208), Amiens, Somme
  - Gustave Roussy-Dermatologie ( Site 1201), Villejuif, Val-de-Marne
  - Hôpital Saint-Louis ( Site 1200), Paris
- Germany (12):
  - Universitätsmedizin Mannheim ( Site 1305), Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Augsburg ( Site 1312), Augsburg, Bavaria
  - Klinik und Poliklinik für Dermatologie und Allergologie-Dermato-oncology ( Site 1315), München, Bavaria
  - Universitätsmedizin Göttingen - Georg-August-Universität-Dermatology ( Site 1308), Göttingen, Lower Saxony
  - Universitätsmedizin Rostock-Klinik und Poliklinik für Dermatologie und Venerologie ( Site 1310), Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum Koeln ( Site 1307), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen-Klinik für Dermatologie, Venerologie und Allergologie ( Site 1300), Essen, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden-Skin Cancer Center Minden ( Site 1301), Minden, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes ( Site 1313), Homburg, Saarland
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien ( Site 1306), Gera, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte-Hauttumorcentrum Charité (HTCC) ( Site 1302), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 1309), Hamburg
- Greece (4):
  - General Hospital of Athens "Laiko"-First Department of Internal Medicine ( Site 3700), Athens, Attica
  - Metropolitan Hospital-A' Oncology Dpt ( Site 3701), Neo Faliro, Attica
  - Bioclinic Thessalonikis Private Clinic Single Member S.A.-Oncology ( Site 3703), Thessaloniki, Central Macedonia
  - European Interbalkan Medical Center-Oncology Department ( Site 3702), Thessaloniki
- Israel (4):
  - Emek Medical Center ( Site 2003), Afula
  - Hadassah Medical Center ( Site 2004), Jerusalem
  - Rabin Medical Center ( Site 2000), Petah Tikva
  - Sheba Medical Center ( Site 2001), Ramat Gan
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1401), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS ( Site 1404), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Senese-U.O.C. Immunoterapia Oncologica ( Site 1402), Siena, Tuscany
  - AO Santa Maria della Misericordia ( Site 1403), Perugia, Umbria
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-s.c. melanoma, immunoterapia oncologica e terapi ( Site 1400), Napoli
- Japan (3):
  - Nagoya University Hospital ( Site 4201), Nagoya, Aichi-ken
  - Shizuoka Cancer Center ( Site 4202), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 4200), Chūō, Tokyo
- New Zealand (2):
  - Capital, Coast and Hutt Valley District - Wellington Regional Hospital ( Site 1502), Newtown, Wellington Region
  - Harbour Cancer & Wellness ( Site 1500), Auckland
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 2909), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2908), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2903), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 2900), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2905), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Chirurgii Onkologicznej, Transplantacyjnej i Ogólnej ( Site 2906), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 2907), Gliwice, Silesian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 2904), Szczecin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Onkologii Klinicznej, Dzial Ch ( Site 2902), Kielce, Świętokrzyskie Voivodeship
- Portugal (4):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil ( Site 3601), Lisbon, Lisbon District
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 3602), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 3603), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 3604), Porto
- South Africa (3):
  - Medical Oncology Centre of Rosebank ( Site 4106), Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 4103), Pretoria, Gauteng
  - Cape Town Oncology Trials ( Site 4100), Cape Town, Western Cape
- South Korea (5):
  - Kyungpook National University Chilgok Hospital-Hematology/oncology ( Site 3904), Daegu, Taegu-Kwangyokshi
  - Chungnam national university hospital-Department of Internal Medicine ( Site 3903), Daejeon, Taejon-Kwangyokshi
  - Seoul National University Hospital-Oncology ( Site 3902), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 3901), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 3900), Seoul
- Spain (6):
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 1600), Barcelona, Catalonia
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 1603), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramón y Cajal ( Site 1602), Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General-Oncology ( Site 1605), Málaga, Malaga
  - HOSPITAL CLINICO DE VALENCIA ( Site 1604), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1601), Barcelona
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 3201), Lund, Skåne County
  - Sahlgrenska Universitetssjukhuset ( Site 3200), Gothenburg, Västra Götaland County
- Switzerland (2):
  - UniversitätsSpital Zürich-Dermatology ( Site 1700), Zürich Flughafen, Canton of Zurich
  - Kantonsspital Graubünden-Medizin ( Site 1703), Chur, Kanton Graubünden
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 4000), Kaohsiung City
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 4004), Tainan
  - National Taiwan University Hospital ( Site 4001), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 4003), Taoyuan District
- Turkey (Türkiye) (7):
  - Hacettepe Universite Hastaneleri ( Site 3006), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 3010), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 3002), Ankara
  - Acibadem Universitesi Atakent Hastanesi-Medical Oncology ( Site 3008), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 3003), Istanbul
  - Ege University Medical Faculty Hospital ( Site 3011), Izmir
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 3005), Izmir
- United Kingdom (9):
  - Bristol Haematology and Oncology Centre ( Site 1811), Bristol, Bristol, City of
  - Addenbrooke's Hospital ( Site 1800), Cambridge, Cambridgeshire
  - Norfolk and Norwich University Hospitals NHS Foundation Trust ( Site 1813), Cringleford, England
  - University College London Hospital ( Site 1807), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 1804), London, London, City of
  - Western General Hospital ( Site 1806), Edinburgh, Midlothian
  - The Churchill Hospital ( Site 1805), Oxford, Oxfordshire
  - St James's University Hospital-Leeds Cancer Centre ( Site 1808), Leeds
  - The Christie NHS Foundation Trust ( Site 1814), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26237&tenant=MT_MSD_9011